CLINICAL TRIAL: NCT03062046
Title: Evaluation of Ablation Index and VISITAG™ Use for Pulmonary Vein Isolation (PVI) in Patients With Paroxysmal Atrial Fibrillation (PAF)
Brief Title: Evaluation of Ablation Index and VISITAG™ (ABI-173)
Acronym: VISTAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-173
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RF ablation (Experimental): Subjects undergoing RF ablation with the Thermocool SmartTouch® (ST) or SmartTouch Surroundflow® (STSF) catheter for treatment of drug resistant symptomatic paroxysmal AF
  Interventions: Device: RF ablation

INTERVENTIONS:
Device: RF ablation — RF ablation

SUMMARY:
The purpose of this study is to assess the safety, acute and long term effectiveness, during standard RF ablation procedures while using Ablation Index and VISITAG™ software in combination with a Thermocool SmartTouch® (ST) or SmartTouch Surroundflow® (STSF) catheter. Furthermore, the role of Ablation Index and VISITAG™ workflow in creating contiguous ablation lines is assessed. The study is a prospective, non-randomized, post-market clinical evaluation. Up to 330 patients will be included in this study. All patients who qualify based on the study specific requirements will be invited to participate. The total duration of the study is estimated to be about 24 months (12 months enrollment period and 12 months of follow up). The clinical investigation population include subjects undergoing RF ablation for treatment of drug resistant symptomatic paroxysmal AF. Prior to enrollment in the clinical investigation, all subjects must meet the inclusion/exclusion criteria and are suitable candidates for enrollment in a clinical investigation in the opinion of the investigator. Subjects must have failed at least one antiarrhythmic drug (AAD) (Type I or III, including β-blocker) as evidenced by recurrent or are intolerant of the AAD.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic paroxysmal AF who had at least one AF episode electrocardiographically documented within one (1) year prior to enrollment. Documentation may include electrocardiogram (ECG); Transtelephonic monitoring (TTM), holter monitor or telemetry strip
2. Failed at least one antiarrhythmic drug (AAD) (Type I or III, including β-blocker) as evidenced by recurrent symptomatic AF, or intolerance to the AAD
3. Age 18 years or older
4. Signed Patient Informed Consent Form (ICF)
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

1. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous LA ablation or surgery
3. Anticipated to receive ablation outside the PV ostia and CTI region
4. Previously diagnosed with persistent AF (> 7 days in duration)
5. LA size >50 mm
6. LA thrombus
7. LVEF < 40%
8. Uncontrolled heart failure or NYHA Class III or IV
9. History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
10. History of a documented thromboembolic event (including TIA) within the past 6 months
11. Previous PCI/MI within the past 3 months
12. Previous cardiac surgery (e.g. CABG) within the past 6 months
13. Previous valvular cardiac surgical/percutaneous procedure (e.g. ventriculotomy, atriomy, valve repair or replacement, presence of a prosthetic valve)
14. Unstable angina pectoris
15. Awaiting cardiac transplantation, cardiac surgery or other major surgery within the next 12 months.
16. Significant pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
17. Acute illness, active systemic infection or sepsis
18. Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
19. Presence of a condition that precludes vascular access
20. Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this trial
21. Current enrollment in an investigational study evaluating another device or drug.
22. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
23. Life expectancy less than 12 months
24. Presenting contra-indications for the devices used in the study, as indicated in the respective Instructions For Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of primary adverse events | 7 days
  A Primary adverse event (PAE) is a serious adverse event, which occurs within the first week (7 days) following an AF ablation procedure with use of ablation index.
confirmation of entrance block | intraoperative
  Presence/absence of acute reconnection will be evaluated through a 30 minute waiting period and adenosine challenge. PVs where acute reconnection is identified during the waiting period or following adenosine challenge will be considered ablation index false positives
long-term effectiveness | 12 months
  Freedom from documented atrial arrhythmia (atrial fibrillation (AF), atrial tachycardia (AT) or atrial flutter (AFL)) episodes (episodes ≥ 30 sec on arrhythmia monitoring device) during the effectiveness evaluation period (day 91-365)

SECONDARY OUTCOMES:
Incidence of individual PAE versus total number of PAE | 12 months
  Incidence of individual PAE versus total number of PAE occured during study
Incidence of entrance block after first encirclement (prior to 30-min waiting period) | intraoperative
  % of subjects with ipsilateral PV isolation (entrance block) after first encirclement (evaluated prior to the 30 minute waiting period and adenosine challenge)
Long-term effectiveness: freedom from documented symptomatic atrial arrhythmia | from 3 up to 12 months
  Freedom from documented symptomatic atrial arrhythmia (AF, AT and AFL) episodes (episodes ≥ 30 sec on arrhythmia monitoring device) during the effectiveness evaluation period (day 91-365)

CONTACTS AND LOCATIONS:
Locations (17):
- LKH Univ. Klinikum Graz, Graz, Austria
- Belgium (4):
  - OLV Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - ZOL Genk, Genk
  - Jessa Ziekenhuis, Hasselt
- Denmark (3):
  - Aarhus Universitetshospital Skejby, Aarhus
  - Gentofte Hospital, Gentofte Municipality
  - Odense University Hospital, Odense
- France (2):
  - Clinique Clairval Marseille, Marseille
  - Clinique Pasteur, Toulouse
- Mater Private Heart & Vascular Centre, Dublin, Ireland
- Italy (2):
  - Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Caisilino Roma, Rome
- Medisch Spectrum Twente, Enschede, Netherlands
- Herzzentrum, Luzerner Kantonsspital, Lucerne, Switzerland
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gupta D, Vijgen J, Potter T, Scherr D, Van Herendael H, Knecht S, Kobza R, Berte B, Sandgaard N, Albenque JP, Szeplaki G, Stevenhagen Y, Taghji P, Wright M, Duytschaever M. Quality of life and healthcare utilisation improvements after atrial fibrillation ablation. Heart. 2021 Aug;107(16):1296-1302. doi: 10.1136/heartjnl-2020-318676. Epub 2021 May 5. PMID 33952593
- [Derived] Duytschaever M, Vijgen J, De Potter T, Scherr D, Van Herendael H, Knecht S, Kobza R, Berte B, Sandgaard N, Albenque JP, Szeplaki G, Stevenhagen YJ, Taghji P, Wright M, Macours N, Gupta D. Standardized pulmonary vein isolation workflow to enclose veins with contiguous lesions: the multicentre VISTAX trial. Europace. 2020 Nov 1;22(11):1645-1652. doi: 10.1093/europace/euaa157. PMID 32879974